CLINICAL TRIAL: NCT01835938
Title: Dose Finding and Early Efficacy Study of Erlotinib in Treatment of Chronic Hepatitis C Virus infection_proof of Concept Study
Brief Title: Clinical Investigation of Erlotinib as an HCV Entry Inhibitor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 5189
Record Dates: First submitted 2013-04-09; First posted 2013-04-19 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Hepatitis C Infection; HCV Genotype 1b
Keywords: Hepatitis C Virus infection; entry inhibitor; kinase inhibitor
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1- Erlotinib (Experimental): Erlotinib is a first class HCV entry inhibitor. In this study, Erlotinib will be administered in escalating doses in sequential patient cohorts for 14 days as follows:
  * Dose level (DL) 1 = 50 mg / day,
  * Dose level (DL) 2 = 100 mg / day, and
  * Dose level (DL) 3 = 150 mg / day .
  Each Dose Level (DL) includes 4 patients (3 patients treated with Erlotinib and one patient treated with the Placebo). Dose escalation will proceed to the subsequent DL in the absence of DLT (dose-limiting toxicity) in 2 patients receiving Erlotinib.
  Interventions: Drug: 1- Erlotinib
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 1- Erlotinib — * Erlotinib 50 mg tablet by mouth every day for 14 days,
  * Erlotinib 100 mg tablet by mouth every day for 14 days,
  * Erlotinib 150 mg tablet by mouth every day for 14 days,
  Arms: 1- Erlotinib
Drug: placebo — * Placebo 50 mg tablet by mouth every day for 14 days,
  * Placebo 100 mg tablet by mouth every day for 14 days,
  * Placebo 150 mg tablet by mouth every day for 14 days,
  Arms: placebo

SUMMARY:
Chronic Hepatitis C Virus (HCV) infection is a major cause of liver cirrhosis and hepatocellular carcinoma world-wide. Current combination therapy of pegylated interferon-alfa, ribavirin and protease inhibitors is limited by resistance and substantial side effects.

The investigators identified epidermal growth factor receptor (EGFR) as host factor for HCV infection. Inhibition of kinase function of EGFR by approved inhibitor Erlotinib (TarcevaTM) broadly inhibits HCV infection of all major genotypes including viral escape variants resistant to host immune responses.

Completed preclinical proof-of-concept studies in HCV cell culture and animal model systems demonstrate that inhibition of EGFR function by Erlotinib constitutes a novel antiviral approach for prevention and treatment of HCV infection (European patent application EP 08 305 604.4, Filing date: September 26, 2008; Inserm, Paris, France and Lupberger et al. Nature Medicine 2011).

Since Erlotinib (TarcevaTM) is an established approved drug for cancer treatment and has a well characterized safety profile in humans, the aim of the study is to investigate the safety, efficacy and pharmacokinetics of Erlotinib, a first-in-class entry inhibitor, for treatment of HCV infection in a randomized placebo-controlled double blind clinical trial in patients chronically infected with HCV. Following completion, this trial will set the stage for a further investigation of entry inhibitors as antivirals in combination with standard of care or direct antivirals such as HCV protease inhibitors. Thus, this randomized clinical trial will be an important step in the development of novel urgently needed antiviral therapies overcoming resistance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic genotype 1b hepatitis C infection with detectable HCV RNA (> 1x104 UI/mL)
* Naïve, relapser or non-responder to interferon with or without ribavirin
* Weight > 45kg, BMI between 18 and 25 Kg/m2 who had a liver biopsy or liver FibroScan eliminating the presence of cirrhosis in the year before enrollment,
* Non-smoker or occasional smoker ( ie < 3 cig/day)

Exclusion Criteria:

* HIV or HBV infection
* Cirrhosis or Liver decompensation
* Chronic liver disease non related to HCV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of virologic response and short-term safety of Erlotinib in patients infected with HCV genotype 1b | 14-day assessment study
  Determination of the recommended dose on the end point of dise-limiting toxicity (DLT), establishment of the maximum-tolerated dose (MTD), and response rate defined as a reduction of at least 1 log10 HCV RNA Levels after the last dose of study drug.

SECONDARY OUTCOMES:
Assessment of pharmacokinetics of Erlotinib in HCV-infected patients | 14-day assessment study
  - Evaluate the pharmacokinetics (AUC, Cmax) of Erlotinib.

OTHER OUTCOMES:
Assessment of Erlotinib in HCV-infected patients and evaluation of drug resistance | 14-day assessment study
  Analyzing the variability of viral species during treatment and evaluate potential resistance to Erlotinib

CONTACTS AND LOCATIONS:
Overall Officials: Dr Samira Fafi-Kremer, Pharma D, PhD, Study Director — Laboratoire de Virologie PTM- Nouvel Hôpital CivilHôpitaux Universitaires de Strasbourg; Dr Catherine Mutter, MD, Study Chair — Centre d'investigation Clinique -P1002Nouvel Hôpital CivilHôpitaux Universitaires de Strasbourg; Dr François Habersetzer, MD, PhD, Study Chair — Service d'Hépato-Gastro-Entérologie - Nouvel Hôpital CivilHôpitaux Universitaires de Strasbourg; Dr. Thomas BAUMERT, MD, PhD, Study Director — Service d'Hépatogastroentérologie, NHC1, place de l'hôpital - BP n°42667091 STRASBOURG CEDEX
Locations (1):
- Service d'Hépatogastroentérologie, NHC1, place de l'hôpital, Strasbourg, Alsace, France